CLINICAL TRIAL: NCT06514716
Title: Role of Intra-articular Corticosteroid Injection in Geniculate Artery Embolization for Knee Osteoarthritis: A Comparative Study
Brief Title: Intra-articular Corticosteroid Injection in GAE for Knee Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed Awad Bessar, Assistant Professor of Diagnostic and Interventional Radiology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GAEIACI-OA
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthritis; Pain, Musculoskeletal
Keywords: Geniculate Artery Embolization; Intra-articular Corticosteroid Injection; Pain Relief; Functional Improvement
MeSH Terms: conditions — Osteoarthritis, Knee; Musculoskeletal Pain | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two groups: Group A receiving geniculate artery embolization (GAE) with intra-articular corticosteroid injection (IACI) and Group B receiving GAE alone.
Who Masked: Outcomes Assessor
Masking Description: Given the specific nature of the interventions, it may not be possible to blind participants or operators; however, to minimize potential bias, outcome assessors will be blinded to the treatment assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GAE with IACI (Experimental): Participants in this arm will undergo geniculate artery embolization (GAE) followed by an intraoperative intra-articular corticosteroid injection (IACI). The procedure aims to alleviate post-procedural pain and improve early functional outcomes in patients with knee osteoarthritis (OA).
  Interventions: Procedure: Geniculate Artery Embolization with Intra-articular Corticosteroid Injection (GAE with IACI)
- GAE alone (Active Comparator): Participants in this arm will undergo geniculate artery embolization (GAE) without the additional intraoperative intra-articular corticosteroid injection. This group will serve as the control to evaluate the effectiveness and safety of GAE with IACI in comparison.
  Interventions: Procedure: Geniculate Artery Embolization alone (GAE alone)

INTERVENTIONS:
Procedure: Geniculate Artery Embolization with Intra-articular Corticosteroid Injection (GAE with IACI) — Participants will undergo geniculate artery embolization (GAE) followed by an intraoperative intra-articular corticosteroid injection (IACI). This combination aims to alleviate post-procedural pain and improve early functional outcomes in patients with knee osteoarthritis (OA).
  Arms: GAE with IACI
Procedure: Geniculate Artery Embolization alone (GAE alone) — Participants will undergo geniculate artery embolization (GAE) without the additional intraoperative intra-articular corticosteroid injection. This procedure aims to serve as a control to evaluate the effectiveness and safety of GAE with IACI in comparison.
  Arms: GAE alone

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness and safety of intra-articular corticosteroid injection (IACI) in alleviating post-procedural pain and improving early outcomes in patients undergoing geniculate artery embolization (GAE) for knee osteoarthritis (OA). The main questions it aims to answer are:

* Does intra-articular corticosteroid injection reduce pain levels post-procedure compared to GAE alone?
* Does the combination of GAE and IACI improve functional outcomes and patient-reported outcomes compared to GAE alone?

Investigators will compare patients receiving GAE with IACI to those receiving GAE alone to see if the addition of IACI provides superior pain relief and functional improvement.

Participants will:

* Undergo geniculate artery embolization, with or without intra-articular corticosteroid injection.
* Have their pain levels assessed using the Visual Analog Scale (VAS) at 1 week, 2 weeks, and 4 weeks post-procedure.
* Complete functional outcome assessments using the KOOS and WOMAC scores.
* Report any adverse events throughout the study period.

DETAILED DESCRIPTION:
This study is a prospective, randomized, comparative trial designed to evaluate the role of intra-articular corticosteroid injection (IACI) in patients undergoing geniculate artery embolization (GAE) for knee osteoarthritis (OA). The trial will enroll adult participants diagnosed with knee OA who are eligible for GAE.

Participants will be randomized into two groups: Group A (GAE with IACI) and Group B (GAE alone). The primary outcome measure will be the Visual Analog Scale (VAS) pain scores at 1 week, 2 weeks, and 4 weeks post-procedure. Secondary outcome measures will include functional improvement assessed using the Knee Injury and Osteoarthritis Outcome Score (KOOS) and the Western Ontario and McMaster Universities Arthritis Index (WOMAC), patient-reported outcomes, and the incidence of adverse events.

The study aims to determine whether the addition of IACI to GAE provides better pain relief and functional outcomes compared to GAE alone. Data will be collected at baseline and specified time points post-procedure, and statistical analysis will be conducted to compare the outcomes between the two groups. This study is conducted in accordance with the principles of the Declaration of Helsinki and has received ethical approval from the institutional review board. Informed consent will be obtained from all participants before enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Diagnosed with knee osteoarthritis (OA) based on clinical and radiographic criteria.
* Eligible for geniculate artery embolization (GAE) as determined by the treating physician.
* Able to provide informed consent and comply with the study protocol.

Exclusion Criteria:

* Contraindications to corticosteroid injections or geniculate artery embolization.
* Pregnant or breastfeeding women.
* Active infection or skin condition at the injection site.
* Severe cardiovascular, renal, or hepatic diseases that may affect study participation.
* Previous knee surgery within the last 6 months.
* Participation in another clinical trial within the last 30 days.
* Inability to comply with follow-up visits or complete study assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-29 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity | 1 week, 2 weeks, and 4 weeks post-procedure
  Pain intensity will be measured using the Visual Analog Scale (VAS) at baseline, 1 week, 2 weeks, and 4 weeks post-procedure.

SECONDARY OUTCOMES:
Functional Improvement (KOOS) | 1 week, 2 weeks, and 4 weeks post-procedure
  Functional improvement will be assessed using the Knee Injury and Osteoarthritis Outcome Score (KOOS) at 1 week, 2 weeks, and 4 weeks post-procedure.
Functional Improvement (WOMAC) | 1 week, 2 weeks, and 4 weeks post-procedure
  Functional improvement will be assessed using the Western Ontario and McMaster Universities Arthritis Index (WOMAC) at 1 week, 2 weeks, and 4 weeks post-procedure.
Incidence of Procedure-Related Adverse Events | Throughout the study period
  Monitoring and recording any adverse events related to the genicular nerve ablation procedures
Patient Satisfaction with the Procedure | 4 weeks post-procedure
  Measured using a structured patient satisfaction questionnaire (PSQ) to gauge participants' satisfaction with the pain relief and overall experience of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Bessar, MD, PhD, Principal Investigator — Assistant Professor of Diagnostic and Interventional Radiology, Zagazig Uni.
Locations (1):
- Zagazig University, Faculty of Medicine, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share individual participant data (IPD) with other researchers. This decision is based on considerations related to patient confidentiality, data privacy concerns, and the absence of a current infrastructure for secure data sharing. The primary results of the study will be published in peer-reviewed journals and presented at scientific conferences, ensuring that the findings are accessible to the broader research community.